CLINICAL TRIAL: NCT03031106
Title: Multidisciplinary Follow-up of Patients Treated for Malignant Hematological Disease; Focus on the Patient's Preferences and Life Situation
Brief Title: Multidisciplinary Follow-up of Patients Treated for Malignant Hematological Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Mia Sommer, Clinical Research Nurse, ph.d. student, Aalborg University Hospital
Other Study IDs: TVO
Record Dates: First submitted 2017-01-12; First posted 2017-01-25 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Malignant Hematologic Neoplasm
Keywords: Patient-reported outcomes, Health-related QoL, Internet-based tool
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to adjust and test an existing internet-based tool for collecting patient-reported outcome measures and to use the internet-based tool in an multidisciplinary follow-up of patients treated for malignant hematological diseases. The patient-reported outcome measurements will be used in describing the patients' health-related quality of life (HRQoL) and to investigate whether the HRQol will increase due to participation in multidisciplinary follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with malignant hematological disease; Morbus Hodgkin and B- and T-cell disease
* patients followed before or after 1. line treatment
* patients in stable phase > 6 months after 1. line treatment
* the patients participation in the study must be assessed and decided by the doctor responsible for the patient's course of treatment

Exclusion Criteria:

* Health conditions which demands close medical monitoring
* conditions which compromise the ability to understand the study and submit informed consent (ex.: dementia and severe mental illness / disability)
* lack of capability to fill out electronic questionnaires
* poor self-care and/or compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with chemotherapy for primary hematological disease and patients followed in a Wait & Watch regimen
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HRQoL) - General | HRQoL is assessed every 2, 3, 4 or 6 months, up to 18 months.
  Patients will be asked to electronically fill out questionnaires before each consultation.
  The questionnaire that will be used to measure HRQoL is SF-36. SF-36 is a generic questionnaire which can be used to assess HRQoL in the general public.
Health-Related Quality of Life (HRQoL) - Disease specific | HRQoL is assessed every 2, 3, 4 or 6 months, up to 18 months.
  Patients will be asked to electronically fill out questionnaires before each consultation.
  The questionnaire that will be used to measure HRQoL is EORTC C30 QLQ. EORTC C30 QLQ is a disease specific questionnaire which can be used to assess HRQoL in patients diagnosed with cancer

SECONDARY OUTCOMES:
Symptoms of depression and anxiety | Symptoms of depression and anxiety will be assessed every 2, 3, 4 or 6 month, up to 18 months
  Data on symptoms of depression and anxiety will be collected before and after each consultation using an international validated questionnaire.
  The questionnaire which will be used is:
  Hospital Depression and Anxiety Scale (HADS)
Symptoms of hematological disease | Symptoms of disease will be assessed every 2, 3, 4 or 6 month, up to 18 months
  Data on symptoms of disease will be collected before each consultation using an international validated questionnaire.
  The questionnaire which will be used is:
  Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF)

CONTACTS AND LOCATIONS:
Overall Officials: Mia Sommer, MHSc, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Department of Hematology, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided